CLINICAL TRIAL: NCT05309278
Title: Effects of a Remote Physical Training Program Combined With Cognitive Training in Older Adults at Increased Risk of Clinical-functional Vulnerability: a Randomized Clinical Trial
Brief Title: Remote Physical and Cognitive Training Effects in Older Adults at Increased Risk of Clinical-functional Vulnerability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Cristine Lima Alberton, Principal investigator, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 55791522.6.0000.5313
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2022-08

CONDITIONS: Aging; Functional Status
Keywords: Exercise; Cognitive training; Aging; Frailty; Occupational performance
MeSH Terms: conditions — Motor Activity; Frailty | interventions — Physical Conditioning, Human; Cognitive Training

STUDY DESIGN:
Intervention Model Description: This is a randomized, single-blind, parallel, controlled, superiority trial. Older participants will be allocated into two groups, experimental and control, based on a randomization sequence that will be generated on a computer in a 1:1 ratio.
Who Masked: Outcomes Assessor
Masking Description: Blinding will be implemented for the outcome assessors. Specifically, all tests, assessments, and measurements will be performed by an investigator blinded to the group participants were assigned to. Because of the type of intervention (i.e., exercise intervention), the investigator(s) who will carry out the exercise sessions, as well as the participants, won't be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical and cognitive exercise group (Experimental): Participants will be randomized to receive physical and cognitive training for a period of 12 weeks.
  Interventions: Behavioral: Physical training; Behavioral: Cognitive training
- Physical exercise only group (Active Comparator): Participants will be randomized to receive only physical training for a period of 12 weeks.
  Interventions: Behavioral: Physical training

INTERVENTIONS:
Behavioral: Physical training — Older adults assigned to this group will undergo two weekly sessions of remote and supervised physical training at home for 1 hour on non-consecutive days. All synchronous meetings will be held on Google Meet, and supervisors will undergo training to standardize their procedures
Behavioral: Cognitive training — These participants will also perform a weekly remote and supervised cognitive training session with neurobic exercises for 1 hour. In addition to the supervised cognitive training session, participants will also be prescribed asynchronous neurobic exercises to be performed on the remaining days of the week (without supervision). The intervention will last for 12 weeks, and all asynchronous neurobic exercises will be recorded in the following synchronous sessions by the supervisor. All synchronous meetings will be held on Google Meet, and supervisors will undergo training to standardize their procedures
  Arms: Physical and cognitive exercise group

SUMMARY:
This study is a randomized, single-blind, parallel, controlled, superiority trial. The main objective is to verify the chronic effects of a remote 12-week low-intensity physical training program alone or in combination with cognitive training on functional, cognitive, and occupational capacity, as well as on the self-reported quality of life.

DETAILED DESCRIPTION:
Participants over 60 years of age at increased risk of clinical-functional vulnerability will be recruited in the city of Pelotas/RS, Brazil and randomized to two different arms. The intervention group will receive low-intensity physical training combined with a cognitive training program using neurobic exercises, whereas the active comparator group will only receive the low-intensity physical training program. Participants from both groups will perform their training sessions remotely for a total of 12 weeks. Outcomes of interest include handgrip strength, functional and cognitive capacity, occupational performance, clinical-functional vulnerability level, self-reported quality of life, and depressive symptoms, which will be assessed in a pre-post fashion. The study hypothesis is that remote low-intensity physical training combined with cognitive training will result in additional benefits to those of low-intensity physical training alone in the physical and cognitive capacity outcomes, and as a consequence, improved quality of life, occupational performance, decreased level of clinical-functional vulnerability and symptoms of depression will be observed.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older,
* MMSE score equal to or greater than 19 points,
* Elementary school education complete or over,
* Sedentary (no current or previous participation in structured exercise (>1x/week) in the past 6 months),
* Increased risk of clinical-functional vulnerability, as determined by the Clinical-Functional Vulnerability Index-20 (IVCF-20) questionnaire.
* Access to a cell phone or notebook with internet access,
* Resident in the city of Pelotas, Brazil.

Exclusion Criteria:

* Individuals who have been affected by COVID-19,
* Not retired, or those retired individuals who maintained continuous or sporadic work activities,
* Neuromuscular deficits or any medical diagnosis that prevents the individuals from performing physical exercises,
* Individuals with decompensated or untreated blood pressure (> than 140x90 mmHg) and,
* Individuals with visual problems that prevent them from watching the training sessions on their cell phone or notebook screen.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) performance | Baseline (weeks 0) to Post-training (week 13)
  The TUG test will be used to measure possible modifications in the dynamic balance of older adults during the performance of the task.
Dual-task performance | Baseline (weeks 0) to Post-training (week 13)
  The TUG test will also be applied with a dual task, in which participants' functional capacity will be assessed while simultaneously performing a verbal task. Specifically, the participants will perform the same procedures explained in the TUG test session, while also pronouncing the maximal number of animal names as possible.
Mini-Mental State Examination (MMSE) score | Baseline (weeks 0) to Post-training (week 13)
  The MMSE will be used to assess participants' cognitive function, which will be classified based on the education-adjusted cut-off scores.

SECONDARY OUTCOMES:
Handgrip strength | Baseline (weeks 0) to Post-training (week 13)
  The amount of force produced by a maximal isometric contraction of the extrinsic hand muscles of the dominant upper limb will be measured using a hand dynamometer.
30-s Sit-to-Stand test performance | Baseline (weeks 0) to Post-training (week 13)
  Lower limb strength will be assessed using the 30-s Sit-to-Stand test, which involves counting the number of times the participant can stand up completely from the sitting position, with arms crossed over the chest.
World Health Organization Quality of Life-bref (WHOQOL-bref) score | Baseline (weeks 0) to Post-training (week 13)
  The WHOQOL-bref questionnaire covers four domains of quality of life (physical health, psychological health, social relationships, and environment) and will be used to assess self-reported quality of life.
Beck's Depression Inventory (BDI) score | Baseline (weeks 0) to Post-training (week 13)
  The BDI is a self-administered questionnaire covering cognitive, affective, behavioral, and somatic aspects of depression.
Canadian Occupational Performance Measure (COPM) | Baseline (weeks 0) to Post-training (week 13)
  The COPM is a semi-structured interview that uses a typical day as a reference to identify issues in self-care, productivity, and leisure based on the self-reported performance capacity and satisfaction of the patient in occupations the participant need, wants, and/or is expected to do.
Digit Span Test (DST) | Baseline (weeks 0) to Post-training (week 13)
  The DST will be used to evaluate participants' working memory.
Verbal fluency test | Baseline (weeks 0) to Post-training (week 13)
  Participants' verbal fluency will me assessed by asking participants to name as many different animals as they know in one minute.

CONTACTS AND LOCATIONS:
Overall Officials: Cristine L Alberton, PhD, Principal Investigator — Federal University of Pelotas
Locations (1):
- Escola Superior de Educação Física, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berni FC, Kanitz AC, Miranda C, de Oliveira DB, Bergamin M, Bullo V, Schaun GZ, Alberton CL. Effects of a remotely supervised physical training program combined with cognitive training for older individuals at increased risk of clinical-functional vulnerability: study protocol for a randomized clinical trial. Trials. 2023 Aug 21;24(1):547. doi: 10.1186/s13063-023-07567-8. PMID 37599360